CLINICAL TRIAL: NCT05258214
Title: Mulligan Bent Leg Raise Versus Mulligan Traction Straight Leg Raise Versus Neural Mobilization With Conventional Therapy On Pain & Functional Disability In Patient With Lumber Radiculopathy
Brief Title: Mulligan BLR Versus Mulligan TSLR Versus Neural Mobilization n Patient With Lumber Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-FSD-00272
Record Dates: First submitted 2022-02-20; First posted 2022-02-28 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Lumbar Radiculopathy
Keywords: Mulligan Technique; Mulligan Traction; Neural Mobilization; Bent Leg Raise; Randomized Control Trial; Straight Leg Raise; Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single Blinding will be performed in this study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mulligan Bent Leg Raise With Conventional Therapy (Experimental): This group will receive mulligan's bent leg raise with conventional therapy. In a mulligan bent leg lift, the practitioner stands on the side of the supine subject on the couch with minimal hamstring stability. The subject's flexed knee is placed over the therapist's shoulder, and the subject is instructed to force the therapist with his leg before relaxing.
  At this moment, the therapist pushes subject's bent knee as high as possible on the same side as his (therapist's) shoulder. Mulligan's Bent Leg is performed three times.
  The raises took 7 seconds to keep and 5 seconds to relax. And conventional therapy includes ultrasound, lumber strengthening, stretching exercises, stabilizing exercises for 30 minutes.
  Interventions: Other: Mulligan Bent Leg Raise
- Mulligan Traction Straight Leg Raise With Conventional Therapy (Experimental): This group will receive mulligan's traction Straight Leg Raise with conventional therapy. Patients were placed in a supine position on a low couch or the floor and provided the Mulligan traction leg raise with knees bent..
  Mulligan's Traction is repeated three times. Straight Leg Raise was kept for 7 seconds and then relaxed for 5 seconds. Three repetitions of the pain-free Straight Leg Raise traction is performed. And conventional therapy include ultrasound, lumber strengthening, stretching exercises, stabilizing exercises for 30 minutes.
  Interventions: Other: Mulligan Traction Straight Leg Raise
- Neural Mobilization With Conventional Therapy (Experimental): This group will receive neural mobilization with conventional therapy. Straight leg raise movements will be used to trigger sciatic nerve pain during neural mobilization exercises.
  Based on the participant's responses and tolerance, several repetitions may be done.
  The range of motion will be expanded as the symptom increases before the full Straight Leg Raise range is reached.
  The position will be kept for a total of 5 minutes and 30 seconds. Repetition will be carried out. And conventional therapy include ultrasound, lumber strengthening, stretching exercises, stabilizing exercises for 30 minutes.
  Interventions: Other: Neural Mobilization

INTERVENTIONS:
Other: Mulligan Bent Leg Raise — Mulligan's bent leg raise, as well as the extreme Straight Leg Raise, can be used to relieve Low Back Pain. It can be used to treat leg discomfort that is above the knee. Bent Leg Raise methods are used where there is a restricted range of motion in the hip flexion joint, as well as low back pressure with or without referred leg pain.
  Arms: Mulligan Bent Leg Raise With Conventional Therapy
Other: Mulligan Traction Straight Leg Raise — Mulligan traction leg raise exercises are a non-invasive treatment that has been shown to help people with low back pain and reduced hip flexion range. Conservative sciatica therapy focuses on pain relief, but increasing Straight Leg Raise range will help restore normal mobility and reduce the severity of low back disability.
  Arms: Mulligan Traction Straight Leg Raise With Conventional Therapy
Other: Neural Mobilization — These techniques are designed to mobilize a nerve with as little pressure down, resulting in a larger longitudinal excursion than techniques that actually lengthen the nerve bed, such as tensioning procedures.
  Arms: Neural Mobilization With Conventional Therapy

SUMMARY:
The goal of this study is to compare the effectiveness of mulligan traction Straight Leg Raise and mulligan's bent leg rise and neural mobilization to conventional therapies in order to assess which treatment is more successful in treating lumbar radiculopathy-related dysfunction.

DETAILED DESCRIPTION:
After the synopsis is approved, Randomized Control Trial study will be performed at Riphah International University Faisalabad. The patients will be enrolled using a targeted sampling method. Patients would be chosen based on pre-established inclusion and exclusion requirements. For this analysis, a sample size estimate shows that 30 randomly selected male or females (18 yrs - 65 yrs) who match the selection criteria will be needed. A basic random sample of 30 lumbar radiculopathy patients was used in an experimental trial. They were divided into three groups of ten people: Group A received neural mobilization with conventional therapy, Group B received mulligan's bent leg rise with conventional therapy, and Group C received mulligan's traction Straight Leg Raise with conventional therapy for six months. Numeric Pain Rating Scale, passive Straight Leg Raise, Goniometer, and modified Oswestry low back pain Questionnaire will be used as outcome tests. After the sixth week, the pre-treatment and post-treatment results will be compared. Each patient will be asked to give their informed consent. Statistical Package of Social Sciences Version 20 can be used for data entry and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65, all genders
* positive slump measure of lumbar specific nerve bias,
* mild to moderate irritation on a Numeric Pain Level Scale of less than seven,
* unilateral radiculopathy in the distribution of a single nerve with a favourable SLR,
* prone knee bent test; positve test,
* hypoaesthesia in a specific dermatome of the unilateral lower limb, accompanied by reduced mobility
* the result of the deep tendon (knee jerk, ankle jerk).

Exclusion Criteria:

* individuals with gradually occurring neurological problems
* Trauma, cancer, and constitutional symptoms are indeed red flags (Fever, Malaise, Weight Loss).
* Hip and knee fractures are common.
* Lower-extremity dislocations.
* Hamstring strains.
* Joint hypermobility of the lower limb.
* Muscle imbalance in lower limb
* Nerve lesions in the lower extremity.
* Subjects who have had low back pain in the previous two months.
* Hip flexion ROM was greater than 100 degrees for the straight knee.
* Neurological defects.
* Metal bolts, plates, or screws in the femur.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 12th Week
  The Numerical Pain Rating Scale is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0; no pain at all to 10; worst imaginable pain.
Modified Oswestry low back pain questionnaire | 12th Week
  Modified Oswestry low back pain questionnaire is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools
Goniometer | 12th Week
  Goniometer has been the most widely used tool for measuring joint range of motion. To ensure reliable measurement, standardized, specific positions and landmarks are used to measure each joint movement.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No